CLINICAL TRIAL: NCT05555966
Title: Electrical Activation Mapping Guided Tailor Made Approach for Cardiac Resynchronization Therapy
Brief Title: CardioInsight 1 RBBB
Acronym: CardioInsight1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Bryan Ping Yen YAN, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017.316
Record Dates: First submitted 2022-09-15; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tailor-made CRT delivery (Experimental): Device placement based on Electrical Activation Mapping result
  Interventions: Device: Electrical Activation Mapping Guided Cardiac resynchronization therapy

INTERVENTIONS:
Device: Electrical Activation Mapping Guided Cardiac resynchronization therapy — To study the feasibility to optimize configuration of CRT delivery for acute correction of electrical dyssynchrony using a noninvasive mapping of global electrical activation

SUMMARY:
Cardiac resynchronization therapy (CRT) is an established therapy for symptomatic heart failure patients. However, there are still 30 to 40% of studied patients being nonresponder to CRT. The plausible reasons of lack of effect of CRT in these patients include relative less baseline electrical dyssynchrony. The aim of our study is to investigate whether there is an optimal configuration of CRT delivery that varies between patients with different pattern of activation delay.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged 18 or above) of both sexes
* Ischemic or non-ischemic cause of heart failure
* QRS duration > 120 ms, non-left bundle branch block (LBBB) type of conduction disturbance
* NYHA class III or above
* Informed consent by the patient
* Already received stable dose of guideline directed medical therapy for at least 3 months

Exclusion Criteria:

* LBBB patients
* Pregnant women
* Participation in another study
* Patient with contraindication to left ventricle catheterization by a retrograde aortic approach

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Left Ventricle (LV) end systolic volume reduction | 6 months
  The responder rate of greater than 10% of LV end systolic volume reduction measured by echocardiogram

SECONDARY OUTCOMES:
Electrical dyssynchrony index | During procedure
  The acute electrical dyssynchrony indices (the standard deviation of activation times throughout the epicardium) of different methods of CRT delivery. Lower indicate larger improvement.
Hemodynamic response monitoring | During procedure
  monitor the difference in hemodynamic responses of different methods of CRT delivery method. The hemodynamic response will be maximal dp/dt as measured by pressure wire introduced into the left ventricle during the procedure.
Procedure outcome with optimal CRT delivery | During procedure
  Procedure outcome measured by procedure duration and implantation success rate of the optimal CRT delivery method as determined by the best improvement in electrical dyssynchrony indices.
Cine images and chest X ray | 6 months
  Cine images (PA, LAO 300, RAO 300) and Chest X ray (PA view) of patients will be obtained for evaluation of changes in disease
Echocardiogram parameter: left ventricular systolic and diastolic volume | 6 months
  left ventricular systolic and diastolic volume at baseline, 3 months and 6 months : , left ventricular ejection fraction, degree of mitral regurgitation, strain imaging will be aggregated to arrive at an overall change in echocardiogram parameters as together they represent integrated heart function collectively, as reflected by the listed echocardiogram parameters.
Multi-dimensional Quality of life changes | 6 months
  change in New York Heart Association (NYHA) class, 6 minute hall walk test, HF Patient Global Assessment Questionnaire and quality of life using Minnesota's living with heart failure (MLWHF) questionnaire at baseline, 3 months and 6 months.
Device set-up parameter :defibrillation threshold | 6 months
  Device parameters including defibrillation threshold at implant and 6 months follow-up.
Post-operation Complication rate | 6 months
  Peri-operative and 6 months follow-up complications rate:
  1. Thromboembolic event
  2. Dislodgement and migration of pacing leads
  3. Phrenic nerve stimulation
  4. Others
Device set-up parameter :defibrillation sensitivity | 6 months
  Device set-up parameter :defibrillation sensitivity at implant and 6 months follow-up
Device set-up parameter: lead impedance of pacing leads | 6 months
  Device set-up parameter: lead impedance of pacing leads at implant and 6 months follow-up
Change in 6 minute hall walk test | 6 months
  Change in 6 minute hall walk test result, at baseline, 3 months and 6 months.
Change in HF Patient Global Assessment Questionnaire | 6 months
  HF Patient Global Assessment Questionnaire at baseline, 3 months and 6 months.
Change in quality of life | 6 months
  Change in quality of life assessed by Minnesota's living with heart failure (MLWHF) questionnaire at baseline, 3 months and 6 months.
Implantation success rate with optimal CRT delivery | During procedure
  Implantation success rate of the optimal CRT delivery method as determined by the best improvement in electrical dyssynchrony indices.
Echocardiogram parameter: left ventricular ejection fraction | 6 months
  Echocardiogram parameter: left ventricular ejection fraction at baseline, 3 months and 6 months
Echocardiogram parameter: degree of mitral regurgitation | 6 months
  Echocardiogram parameter: degree of mitral regurgitation at baseline, 3 months and 6 months
Echocardiogram parameter: strain imaging | 6 months
  Echocardiogram parameter: strain imaging at baseline, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Yan, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong